CLINICAL TRIAL: NCT04879498
Title: Clinical Evaluation of Monolithic Zirconia and Metal-ceramic Posterior Fixed Partial Dentures
Brief Title: Clinical Evaluation of Monolithic Zirconia FPDs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Ivoclar Vivadent AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4155858 Ivoclar Vivadent AG; 15/236-E (Other: Ethical Committee of Clinical Research. Hospital S. Carlos.)
Record Dates: First submitted 2021-04-15; First posted 2021-05-10 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Dental Materials
Keywords: fixed partial dentures; clinical evaluation; monolithic zirconia; veneered zirconia; survival
MeSH Terms: interventions — Metal Ceramic Alloys

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Monolithic zirconia (Experimental): Monolithic zirconia posterior 3-unit fixed partial dentures
  Interventions: Drug: Monolithic zirconia
- Veneered zirconia (Active Comparator): Veneered zirconia posterior 3-unit fixed partial dentures
  Interventions: Other: Veneered zirconia
- Metal-ceramic (Active Comparator): Metal-ceramic posterior 3-unit fixed partial dentures
  Interventions: Other: Metal-ceramic

INTERVENTIONS:
Drug: Monolithic zirconia — To assess the clinical performance and survival of posterior monolithic zirconia fixed partial dentures
  Other Names: Zenostar T; Wieland Dental
  Arms: Monolithic zirconia
Other: Veneered zirconia — To assess the clinical performance and survival of posterior veneered zirconia fixed partial dentures
  Other Names: IPS e.max ZirCAD
  Arms: Veneered zirconia
Other: Metal-ceramic — To assess the clinical performance and survival of posterior metal-ceramic fixed partial dentures
  Arms: Metal-ceramic

SUMMARY:
The objectives of the present study are to compare the survival rates and possible biological and technical complications of metal-ceramic, veneered and monolithic zirconia posterior three-unit fixed partial dentures. The null hypothesis is that no differences would be found between the parameters studied for each type of restoration.

DETAILED DESCRIPTION:
Ninety patients requiring at least one 3-unit Fixed partial denture (FPD) in the posterior region of the maxilla or mandible were included in this study. All subjects were recruited from the Master in Buccofacial Prostheses and Occlusion (Faculty of Odontology, University Complutense of Madrid, Spain). Before treatment, patients were informed of the study objectives, clinical procedures, materials used, advantages and possible risks of the ceramic material, and other therapeutic alternatives. Prior to the study, participants were asked to provide written informed consent. Ninety posterior FPDs were produced and allocated in parallel and randomly to either monolithic zirconia, veneered zirconia or MC restorations. The clinical procedures were performed by two experienced clinicians. All participants received oral hygiene instructions and a professional tooth cleaning prior to prosthetic treatment. The abutment teeth were prepared with a 0.8- to 1-mm-wide circumferential chamfer, an axial reduction of 1 mm and an occlusal reduction of 1.5- to 2.0-mm. A 10- to 15- degree angle of convergence was achieved for the axial walls. Tooth preparations were scanned with an intraoral scanner and the FPDs were designed using specific software. The restorations were then cemented using a resin self-adhesive cement. After cementation, occlusal contacts were evaluated, and the adjusted surfaces were polished using a porcelain polishing kit. The 90 FPDs were examined at 1week (baseline),1, 2 and 2 years by 2 researchers who were not involved in the restorative treatment.

ELIGIBILITY:
Inclusion Criteria:

* One posterior tooth (molar or premolar) to be replaced
* Vital abutments or abutments with an adequate endodontic treatment
* Abutment not crowned previously
* Periodontally healthy abutments with no signs of bone resorption or periapical disease
* Adequate occlusogingival height for an appropiate connector area of at least 9 mm2
* Stable occlusion and the presence of natural dentition in the antagonist arch.

Exclusion Criteria:

* Patients who require a Fixed Dental Prosthesis of more than three units
* Patients who present reduced crown length (less than 3 mm occlusogingival heigth)
* Poor oral hygiene, high caries activity, or active periodontal disease

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-01-18 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Quality of restorations at baseline | Baseline
  The quality of the surface and color, anatomical form and marginal integrity was assessed using the California Dental Association's assessment system. Each CDA criterion was ranked on a scale of 1 to 4, where 4 = excellent, 3 = good, 2 = unacceptable (repair), and 1 = unacceptable (replacement).
Quality of restorations at 1 year | 1 year
  The quality of the surface and color, anatomical form and marginal integrity was assessed using the California Dental Association's assessment system. Each CDA criterion was ranked on a scale of 1 to 4, where 4 = excellent, 3 = good, 2 = unacceptable (repair), and 1 = unacceptable (replacement).
Quality of restorations at 2 years | 2 years
  The quality of the surface and color, anatomical form and marginal integrity was assessed using the California Dental Association's assessment system. Each CDA criterion was ranked on a scale of 1 to 4, where 4 = excellent, 3 = good, 2 = unacceptable (repair), and 1 = unacceptable (replacement).ty was assessed
Quality of restorations at 3 years | 3 years
  The quality of the surface and color, anatomical form and marginal integrity was assessed using the California Dental Association's assessment system. Each CDA criterion was ranked on a scale of 1 to 4, where 4 = excellent, 3 = good, 2 = unacceptable (repair), and 1 = unacceptable (replacement).
Plaque Index (PI) at baseline | Baseline
  Plaque Index (PI) of the abutment and control teeth. A score of 0 to 3 was assigned. Higher score means a worse outcome.
Plaque Index (PI) at 1 year | 1 year
  Plaque Index (PI) of the abutment and control teeth. A score of 0 to 3 was assigned. Higher score means a worse outcome.
Plaque Index (PI) at 2 years | 2 years
  Plaque Index (PI) of the abutment and control teeth. A score of 0 to 3 was assigned. Higher score means a worse outcome.
Plaque Index (PI) at 3 years | 3 years
  Plaque Index (PI) of the abutment and control teeth. A score of 0 to 3 was assigned. Higher score means a worse outcome.
Gingival Index (GI) at baseline | Baseline
  Gingival Index (GI) of the abutment and control teeth. A score of 0 to 3 was assigned. Higher score means a worse outcome.
Gingival Index (GI) at 1 year | 1 year
  Gingival Index (GI) of the abutment and control teeth. A score of 0 to 3 was assigned. Higher score means a worse outcome.
Gingival Index (GI) at 2 years | 2 years
  Gingival Index (GI) of the abutment and control teeth. A score of 0 to 3 was assigned. Higher score means a worse outcome.
Gingival Index (GI) at 3 years | 3 years
  Gingival Index (GI) of the abutment and control teeth. A score of 0 to 3 was assigned. Higher score means a worse outcome.
Margin stability at baseline | Baseline
  To assess the gingival margin stability throughout the evaluation period (subgingival, isogingival or supragingival)
Margin stability at 1 year | 1 year
  To assess the gingival margin stability throughout the evaluation period (subgingival, isogingival or supragingival)
Margin stability at 2 years | 2 years
  To assess the gingival margin stability throughout the evaluation period (subgingival, isogingival or supragingival)
Margin stability at 3 years | 3 years
  To assess the gingival margin stability throughout the evaluation period (subgingival, isogingival or supragingival)
Probing depth at baseline | Baseline
  Probing depth of the abutment and control teeth. A score of 0 to 4 was assigned. Higher score means a worse outcome
Probing depth at 1 year | 1 year
  Probing depth of the abutment and control teeth. A score of 0 to 4 was assigned. Higher score means a worse outcome
Probing depth at 2 years | 2 years
  Probing depth of the abutment and control teeth. A score of 0 to 4 was assigned. Higher score means a worse outcome
Probing depth at 3 years | 3 years
  Probing depth of the abutment and control teeth. A score of 0 to 4 was assigned. Higher score means a worse outcome
Patient satisfaction at 3 years | 3 years
  Subjective patient satisfaction using Visual analogue scale (VAS) ranged from 0 (worst possible result) to10 (best possible result). The items analyzed were: esthetics, function, comfort, overall satisfaction